CLINICAL TRIAL: NCT05161676
Title: Modulation of Circulating Levels of the Ketone Body 3-hydroxybutyrate in Patients With Chronic Heart Failure: Metabolic Effects
Brief Title: Metabolic Effects of Chronic Ketosis (KETO-CHF Metabolic)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristoffer Berg-Hansen, MD, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KETO-CHF Metabolic
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (3-OHB) (Experimental)
  Interventions: Dietary Supplement: Ketone monoester
- Placebo Treatment (Experimental)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Commercially available ketone supplement
  Arms: Ketone monoester (3-OHB)
Dietary Supplement: Placebo drink — Isocaloric placebo
  Arms: Placebo Treatment

SUMMARY:
Heart Failure (HF) is a major public health issue because the disease affects 1-2% of the Western population and the lifetime risk of HF is 20%. Despite major improvements in the management and care of patients with HF, the 1-year mortality in patients with HF is 13% and >50% of HF patients are admitted during a 2.5 year period. Furthermore, patients with HF have markedly decreased physical capacity and quality of life. Thus, there is a need for new treatment modalities in this group of patients.

It is well established that patients with heart failure have metabolic disturbances, including disturbed glucose metabolism with increasing insulin resistance, increased lipolysis, and disturbances in skeletal muscle homeostasis.

Presently there are no data on the clinical metabolic effects of long-term oral ketone-supplementation in patients with chronic HF.

In this study we aim to investigate the effect of 14 days modulation of circulating ketone body levels on endogenous protein, glucose, and fatty acid metabolism in patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with NYHA II-III
* Left ventricular ejection fraction ≤40%
* Negative urine-HCG for women with childbearing potential

Exclusion Criteria:

* Known diabetes or HbA1c ≥48 mmol/mol
* Significant cardiac valve disease
* Severe stable angina pectoris
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Differences in lipolysis rate | 14 days of dietary supplement
  Measured as differences in palmitate flux

SECONDARY OUTCOMES:
Changes in protein metabolism | 14 days of dietary supplement
  Measured with a urea tracer
Changes in glucose kinetic | 14 days of dietary supplement
  Measured by glucose tracer

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided